CLINICAL TRIAL: NCT06384300
Title: Financial Incentives and Motivational Intervention to Improve Gastric Cancer Screening in China: An Individual Level Randomized Controlled Trial Study Protocol
Brief Title: Financial Incentives and Motivational Intervention to Improve Gastric Cancer Screening in China
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Li Yang, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BMSF
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Screening; Random Control Trial; China
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (No Intervention): This is the control group.
- Group B (Experimental): In the financial incentive group (Group B), participants will receive reimbursement for transportation, accommodation, and food costs, along with RMB 200 (about 30 US dollar) to compensate for potential income loss due to endoscopy, provided they undergo the procedure.
  Interventions: Other: Financial Incentives
- Group C (Experimental): For the motivational intervention group (Group C), researchers will provide detailed information about the social norms surrounding endoscopy screening, including the prevalence of screening participation, the potential risks of gastric cancer, and the health benefits of screening.
  Interventions: Other: Motivational Intervention
- Group D (Experimental): Participants in the mixed intervention group (Group D) will receive both financial incentives and motivational intervention.
  Interventions: Other: Mixed Intervention

INTERVENTIONS:
Other: Financial Incentives — In the financial incentive group, participants will receive reimbursement for transportation, accommodation, and food costs, along with RMB 200 (about 30 US dollar) to compensate for potential income loss due to endoscopy, provided they undergo the endoscopy.
  Arms: Group B
Other: Motivational Intervention — For the motivational intervention group, researchers will provide detailed information about the social norms surrounding endoscopy screening, including the prevalence of screening participation, the potential risks of gastric cancer, and the health benefits of screening.
  Arms: Group C
Other: Mixed Intervention — Participants in the mixed intervention group will receive both financial incentives and motivational intervention.
  Arms: Group D

SUMMARY:
Gastric cancer, also known as stomach cancer, is a serious disease that affects the stomach. It's one of the most common types of cancer, and sadly, many people die from it each year. But there's hope! We can catch gastric cancer early with a special test called endoscopy. This test helps doctors find cancer or pre-cancerous changes in the stomach early, when it's easier to treat. However, not enough people get this test, especially in places where healthcare isn't easily available. That's why we're doing this study.

We want to find out if we can encourage more people to get the endoscopy test for gastric cancer. We're going to try two different ways to encourage people to get the test. First, we'll give some people money or other incentives to help cover the costs of getting the test. Second, we'll give others information and support to help them understand why the test is important and how it can help them.

We'll be doing this study in two provinces in China, where gastric cancer is a big problem. We'll ask thousands of people to join the study, and we'll randomly assign them to one of the two groups. Then, we'll see if more people in one group get the endoscopy test compared to the other group.

Our hope is that by finding out what works best, we can help more people catch gastric cancer early and get the treatment they need. This could save many lives and make a big difference in fighting this disease.

DETAILED DESCRIPTION:
Gastric cancer (GC) remains a significant global health challenge, with high mortality rates, particularly in low- and middle-income country, like China. Early detection through screening is crucial for improving prognosis and reducing mortality. However, uptake of GC screening remains suboptimal, highlighting the need for effective interventions to promote screening participation.

This study employs an experimental design to evaluate the effectiveness of two interventions, financial incentives and motivational interventions, in promoting GC screening uptake at the individual level. A large sample size will be recruited from high GC-burden provinces in China, and participants will be randomly assigned to intervention and control groups. Statistical analyses, including Propensity Score Matching and Interrupted Time Series Analysis, will be utilized to assess the impact of interventions on screening uptake and adherence.

Findings from this study will be disseminated through peer-reviewed publications, conference presentations, and engagement with stakeholders to inform evidence-based strategies for improving GC screening and reducing GC-related morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent by patients;
2. Identification as "high risk" (≥5 scores) by Gastric Cancer Risk Scoring System (GC-RSS).

Exclusion Criteria:

1. History of previous gastric cancer screening, including endoscopy and serum biomarker examination (pepsinogen, G-17, and MG7-Ag);
2. Diagnosis of cancer or presence of precancerous lesions or conditions;
3. Having family members who have already participated in this study;
4. Diagnosis of severe depression or psychiatric disorder;
5. Presence of other medical conditions that preclude receipt of endoscopy services.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1 | 3 month (90 days)
  Our primary outcome is the rate of individuals undergoing endoscopy screening within three months.
Primary Outcome 2 | 6 month (180 days)
  Our primary outcome is the rate of individuals undergoing endoscopy screening within six months.

SECONDARY OUTCOMES:
Secondary Outcome | 1 or 2 years
  the proportion of participants adhering to follow-up endoscopy appointments at one- or two-years post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, PhD, Study Director — Peking University

IPD SHARING:
Plan to Share IPD: No